CLINICAL TRIAL: NCT01418612
Title: An Open Label, Randomised, Two Period, Two Treatment, Two Sequence, Crossover, Single-Dose Bioequivalence Study of Venlafaxine Hydrochloride Extended-Release Capsules 150mg (Test Formulation, Torrent Pharmaceutical Limited., India) Versus Effexor XR® 150mg Capsule (Reference Formulation, Wyeth Pharmaceuticals Inc., USA) in Healthy Volunteers Under Fed Conditions
Brief Title: Bioequivalence Study of Torrent Pharmaceutical Limited's Venlafaxine Hydrochloride ER Capsules Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Chief Investigator, Torrent Pharmaceuticals Limited
Other Study IDs: PK-08-001
Record Dates: First submitted 2011-08-10; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Healthy

INTERVENTIONS:
Drug: Venlafaxine Hydrochloride Extended-Release Capsules of Torrent Pharmaceuticals Limited

SUMMARY:
Objective:

The Bioequivalence studies were performed to compare the rate and extent of release of the drug substance from the two Capsule formulations containing Venlafaxine Hydrochloride Extended-Release Capsules 150mg of Torrent Pharmaceuticals Limited and the Effexor XR® (Venlafaxine Hydrochloride) Extended-Release Capsules 150mg of Wyeth Pharmaceuticals Inc., USA.

Study Design:

Open Label, Randomised, Two Period, Two Treatment, Two Sequence, Crossover, Single-Dose Bioequivalence Study of Venlafaxine Hydrochloride Extended-Release Capsules 150mg (Test formulation, Torrent Pharmaceutical Limited., India) Versus Effexor XR® 150mg capsule (Reference formulation, Wyeth Pharmaceuticals Inc., USA) in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

(*)The volunteers were excluded from the study based on the following criteria:

* Sex: male.
* Age: 18 - 45 years. .
* Volunteer with BMI of 18-27 (inclusive both) kg/m2 with minimum of 50 kg weight.
* Healthy and willing to participate in the study.
* Volunteer willing to adhere to the protocol requirements and to provide written informed consent.
* Non-smokers or smoker who smokes less than 10 cigarettes per day

Exclusion Criteria:

(*)The volunteers were excluded from the study based on the following criteria:

* Clinically relevant abnormalities in the results of the laboratory screening evaluation.
* Clinically significant abnormal ECG or Chest X-ray.
* Systolic blood pressure less than 100 mm Hg or more than 140 mm Hg and diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
* Pulse rate less than 50/minute or more than 100/minute.
* Oral temperature less than 95°P or more than 98.6°P.
* Respiratory rate less than 12/minute or more than 20/minute
* History of allergy to the test drug or any drug chemically similar to the drug under investigation.
* History of alcohol or drug abuse
* Positive breath alcohol test
* Recent history of kidney or liver dysfunction.
* History of consumption of prescribed medication since last 14 days or OTC medication since last 07 days before beginning of the study.
* Volunteers suffering from any chronic illness such as arthritis, asthma etc.
* History of heart failure.
* HIV, HCV, HBsAg positive volunteers.
* Opiate, tetra hydrocannabinol, amphetamine, barbiturates, benzodiazepines, - Cocaine positive volunteers based on urine test.
* Volunteers suffering from any psychiatric (acute or chronic) illness requiring medications.
* Administration of any study drug in the period 0 to 3 months before entry to the study.
* History of significant blood loss due to any reason, including blood donation in the past 3 months.
* History of pre-existing bleeding disorder.
* Existence of any surgical or medical condition, which, in the judgment of the chief investigator and/or clinical investigator/physician, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of volunteers.
* Inability to communicate or co-operate due to language problem, poor mental development or impaired cerebral function.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult

PRIMARY OUTCOMES:
Bioequivalence based on Composite of Pharmacokinetics
  Bioequivalence; 90% geometric confidence interval of the ratio of least-squares means of the test to reference product should be within 80.00% - 125.00% for AUC-unf, AUCo-t and Cmax.

CONTACTS AND LOCATIONS:
Locations (1):
- Bio Evaluation Centre, Torrent Pharmaceuticals Ltd.,, Village Bhat, Gandhinagar, Gujarat, India